CLINICAL TRIAL: NCT01458067
Title: A Phase I/IIa, First Time in Human, Open-label Dose-escalation Study of GSK2636771 in Subjects With Advanced Solid Tumors With PTEN Deficiency
Brief Title: A Phase I/IIa, First Time in Human, Study of GSK2636771 in Subjects With Advanced Solid Tumors With Phosphatase and Tensin Homolog (PTEN) Deficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115717
Record Dates: First submitted 2011-10-13; First posted 2011-10-24 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — GSK2636771

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 (Experimental): GSK2636771 single dose and then daily dosing after approximately 1 week
  Interventions: Drug: GSK2636771
- Part 2 (Experimental): GSK2636771 single dose and then daily dosing starting on Day 4
  Interventions: Drug: GSK2636771
- Part 3 (Experimental): GSK2636771 daily dosing
  Interventions: Drug: GSK2636771

INTERVENTIONS:
Drug: GSK2636771 — Oral capsules

SUMMARY:
The study consists of a pre-screening period to determine if the subject's tumor has PTEN deficiencies. Subjects then continue into the screening phase for Part 1, 2, or 3, as appropriate. In Part 1, subjects will then receive a single dose of 25 mg. After analysis of 24 hour pharmacokinetic (PK) samples, subjects may receive continuous dosing or receive a single modified dose. In Part 2, subjects will be enrolled and dose escalation will occur in a 3+3 design. Subjects will receive a single dose on Day 1, and then begin continuous daily dosing after collection of a 72-hour PK sample. Additional subjects may be enrolled at lower dose levels for assessment of pharmacodynamic response. In Part 3, up to two tumor-specific expansion cohorts will be enrolled and receive the MTD or BED as defined in Part 2. A minimum of 12 and a maximum of 20 evaluable subjects will be enrolled in each cohort. Interim monitoring for futility will be incorporated after response data from 12 subjects are available. In addition, up to 20 evaluable subjects will be enrolled into Part 3 -Signal-finding Expansion Cohort at the MTD or BED as defined in Part 2. All subjects in all parts/cohorts will receive daily dosing until withdrawal or unacceptable toxicity. All subjects in all parts/cohorts will receive daily dosing until withdrawal or unacceptable toxicity.

DETAILED DESCRIPTION:
The study consists of a pre-screening period to determine if the subject's tumor has PTEN deficiencies. Subjects then continue into the screening phase for Part 1, 2, or 3, as appropriate. In Part 1, subjects will then receive a single dose of 25 mg. After analysis of 24 hour pharmacokinetic (PK) samples, subjects may receive continuous dosing or receive a single modified dose. In Part 2, subjects will be enrolled and dose escalation will occur in a 3+3 design. Subjects will receive a single dose on Day 1, and then begin continuous daily dosing after collection of a 72-hour PK sample. Additional subjects may be enrolled at lower dose levels for assessment of pharmacodynamic response. In Part 3, up to two tumor-specific expansion cohorts will be enrolled and receive the MTD or BED as defined in Part 2. A minimum of 12 and a maximum of 20 evaluable subjects will be enrolled in each cohort. Interim monitoring for futility will be incorporated after response data from 12 subjects are available. In addition, up to 20 evaluable subjects will be enrolled into Part 3 -Signal-finding Expansion Cohort at the MTD or BED as defined in Part 2. All subjects in all parts/cohorts will receive daily dosing until withdrawal or unacceptable toxicity. All subjects in all parts/cohorts will receive daily dosing until withdrawal or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

Pre-screening Parts 1, 2, and 3

* Male or female at least 18 years of age at the time of signing the informed consent form and capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Performance Status score of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
* Able to swallow and retain orally administered medication.
* Sufficient archival tumor biopsy specimen is available for PTEN IHC analysis, or subject is willing to undergo a fresh tumor biopsy for PTEN IHC analysis.

Pre-screening Parts 1 and 2 only

* Histologically or cytologically confirmed diagnosis of one of the following solid tumor malignancies that is not responsive to standard therapies or for which there is no approved or curative therapy or for subjects that refuse standard therapy: Endometrial cancer (endometriod), Prostate cancer, Ovarian cancer, Non-small cell lung cancer, Breast cancer (ER, PR, and HER2 negative), Gastric adenocarcinoma, Colorectal cancer, Head/neck squamous cell carcinoma, Melanoma, or Glioblastoma multiformae at first or second recurrence (more specific disease history is detailed in the study protocol).

Pre-screening Part 3 only

* Must have tumor amenable to biopsy Pre-screening Part 3 CRPC cohort only: prostate adenocarcinoma, surgically castrated or continuously medically castrated (for greater than or equal to 8 weeks prior to pre-screening), and
* persistent disease with evidence of disease progression following standard therapy(ies) including prior treatment with docetaxel and androgen/androgen receptor directed therapy, including enzalutamide and/or abiraterone
* serum testosterone level <1.7 nmol/L or <50 ng/dL
* PSA level of greater than or equal to 2.0 ng/mL For CRC cohort: CRC with persistent disease with evidence of disease progression following standard therapy(ies) that included multi-agent chemotherapy regimen(s) with exposure to oxaliplatin and irinotecan.

For Signal-finding Expansion Cohort: one of the specified tumor types that is not responsive to standard therapies, or for which there is no approved or curative therapy, or for which subjects have refused standard therapy, including:

* Triple negative breast cancer (ER, PR, and HER2 negative), Endometriod, Gastric, Glioblastoma multiformae, Head/neck squamous cell carcinoma, Melanoma, Non-small cell lung cancer, Ovarian Screening Parts 1, 2 includes Pre-screening criteria (above) and
* For Parts 1 and 2, histologically or cytologically confirmed diagnosis of one of the following solid tumor malignancies that is not responsive to standard therapies or for which there is no approved or curative therapy or for subjects that refuse standard therapy: Endometrial cancer (endometriod), Prostate cancer, Ovarian cancer, Non-small cell lung cancer, Breast cancer (ER, PR, and HER2 negative), Gastric adenocarcinoma, Colorectal cancer, Head/neck squamous cell carcinoma, Melanoma, or Glioblastoma multiformae at first or second recurrence (more specific disease history is detailed in the study protocol). For Part 3, histologically or cytologically confirmed diagnosis of one of the following solid tumor malignancies that is not responsive to standard therapies or for which there is no approved or curative therapy or for subjects that refuse standard therapy: Endometrial cancer (endometriod), Prostate cancer, or Gastric adenocarcinoma.
* All prior treatment-related toxicities must be National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0, <=Grade 1 (except alopecia) at the time of treatment allocation with the exception of peripheral neuropathy, which must be <=Grade 2.
* Adequate organ system function defined as ANC greater than or equal to 1X10^9/L without growth factor in the past 7 days, hemoglobin greater than or equal to 9g/dL without transfusion in the past 7 days, platelets greater than or equal to 75X10^9/L without transfusion in the past 7 days, PT/INR and PTT less than or equal to 1.5XULN, total bilirubin less than or equal to 1.5XULN (isolated bilirubin >1.5XULN is acceptable if bilirubin is fractionated and direct bilirubin <35%), AST and ALT less than or equal to 2.5XULN (AST/ALT can be up to 4XULN in the presence of liver metastasis, but cannot be associated with elevated bilirubin), calculated creatinine clearance or 24-hour urine creatinine clearance greater than or equal to 50mL/min, cardiac ejection fraction greater than or equal to LLN by echocardiography.
* Women of childbearing potential and men with reproductive potential must be willing to practice acceptable methods of birth control prior to and after the start of dosing. Additionally, women of childbearing potential must have a negative serum pregnancy test within 14 days prior to the first dose of study medication.
* Subjects must have tumors with a documented PTEN deficiency using an analytically validated IHC assay or other correlative assay (e.g., FISH). Determination of PTEN deficiency using archival tumor is acceptable. Where archival tissue is not available or does not confirm PTEN deficiency, a fresh tumor sample will be acceptable for screening, and those with PTEN deficiency will be eligible.
* Subjects enrolled as part of PD expansion group (Part 2) must agree to undergo pre- and on-treatment tumor biopsies.

Screening Part 3 includes Pre-screening criteria (above) and

* UPC <0.2
* Must continue to have tumor amenable to biopsy
* Must agree to undergo both pre-treatment and on-treatment tumor biopsies
* Male Subjects of Reproductive Potential: Subjects must agree to use effective contraception throughout the treatment period and for five days after the last dose of study treatment.

Exclusion Criteria:

Pre-screening Parts 1, 2, and 3

* Presence of any clinically significant GI abnormalities or other condition that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* History of congenital platelet function defect (e.g., Bernard-Soulier syndrome, Chediak-Higashi syndrome, Glanzmann thrombasthenia, storage pool defect)
* Any serious or unstable pre-existing medical, psychiatric, or other condition (including laboratory abnormalities) that could interfere with subject's safety or providing informed consent.

Screening Parts 1, 2 includes Pre-screening criteria (above) and

* Subject has had chemotherapy, radiotherapy, immunotherapy, or other anti-cancer therapy including investigational drugs within 14 days prior to the first dose of the investigational drug described in this study. Hormonal (e.g., anti-androgen) therapies for prostate cancer must be stopped 4 to 6 weeks prior to enrolment. NOTE: Subjects with prostate cancer may remain on LHRH agonists. Subjects with prostate cancer may remain on low-dose prednisone or prednisolone (up to 10 mg per day) and still be eligible for this study.
* Current use of prohibited medication during treatment with GSK2636771. Current use of aspirin, clopidogrel, ticlopidine, prasugrel, or ticagrelor is prohibited. Anticoagulants are permitted only if the subject meets PTT and INR entry criteria. Their use must be monitored in accordance with local institutional practice.
* Active peptic ulcer disease or history of abdominal fistula, GI perforation, or intra abdominal abscess within 28 days prior to beginning study treatment.
* Any major surgery within the last four weeks.
* Poorly controlled hypertension (defined as systolic blood pressure of >=150 mmHg or diastolic blood pressure of >100 mmHg based on a mean of 3 measurements at approximately 2-minute intervals). NOTE: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry.
* Known active infection requiring parenteral or oral anti-infective treatment.
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal or cardiac disease).
* Subjects with brain metastases of non-central nervous system (CNS) primary tumors are excluded if their brain metastases are:

  * Symptomatic
  * Treated (surgery, radiation therapy) but not clinically and radiographically stable one month after local therapy (as assessed by contrast enhanced magnetic resonance imaging [MRI] or computed tomography [CT]), OR
  * Asymptomatic and untreated but >1 cm in the longest dimension
  * Subjects with small (<=1 cm in the longest dimension), asymptomatic brain metastases that do not need immediate local therapy can be enrolled.
  * NOTE: Subjects on a stable (i.e., unchanged) dose of corticosteroids for more than one month, or those who have been off corticosteroids for at least 2 weeks can be enrolled. Subjects must also be off of enzyme-inducing anticonvulsants for more than 4 weeks
* QTcF interval >=470 msecs. If a screening QTcF is >=470 msecs, it should be repeated 2 additional times at least 5 minutes apart and the average of the 3 readings should be used to determine eligibility.
* Other clinically significant ECG abnormalities including 2nd degree (Type II) or 3rd degree atrioventricular block.
* History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within the past 6 months.
* Class III or IV heart failure as defined by the New York Heart Association functional classification system.
* Baseline cardiac troponin (cT-n) >10% coefficient of variance (CV).
* Known hypersensitivity to any of the components of the study treatment.
* Pregnant or lactating female.
* Any malignancy related to human immunodeficiency virus (HIV) or solid organ transplant; history of known HIV, history of known Hepatitis B virus (HBV) surface antigen positivity (subjects with documented laboratory evidence of HBV clearance may be enrolled) or positive Hepatitis C virus antibody confirmed by recombinant immunoblot assay.

Screening Part 3 includes Pre-screening criteria (above) and

* Prior treatment with: Anti-cancer therapy (e.g., chemotherapy with delayed toxicity,immunotherapy, biologic therapy or chemoradiation) within 21 days (or within 42 days if prior nitrosourea or mitomycin C containing therapy)prior to enrollment and/or daily or weekly chemotherapy without the potential for delayed toxicity within 14 days prior to enrollment • Investigational drug(s) within 30 days or five half-lives, whichever is longer, prior to enrollment
* Current use of prohibited medication(s) or requirement for prohibited medication(s) during study treatment NOTE: Current use of anticoagulants is permitted if the subject meets the PTT and INR entry criteria (see Table 6) and monitored in accordance with local institutional practice. NOTE: Subjects who are currently on an aspirin regimen or using aspirin containing product(s) at the time of screening MUST agree to discontinue aspirin or aspirin-containing product(s) at least 10 days prior to first dose of study treatment. After study Day 22 and completion of all assessments to be performed during this period, including tumor biopsies, the aspirin regimen or use of aspirin-containing product(s) may be resumed CRPC cohort only: subjects may remain on LHRH agonists (i.e., leuprolide, goserelin, triptorelin or histrelin), low dose prednisone or prednisolone (up to 10 mg/day), or bisphosphonates (if on stable dose for at least four weeks) without interruption and remain eligible for this study.
* Any unresolved greater than or equal to Grade 2 (per CTCAE, v 4.0) toxicity from previous anti-cancer therapy, except alopecia or Grade 2 anemia (if hemoglobin is greater than or equal to 9.0 g/dL)
* Any greater than or equal to Grade 3 (per CTCAE, v 4.0) electrolyte abnormality
* Any greater than or equal to Grade 2 (per CTCAE, v 4.0) hypocalcemia (except where ionized calcium is less than or equal to Grade 1), hypokalemia, hyponatremia, hypomagnesemia, or symptomatic hypophosphatemia
* Active peptic ulcer disease or history of abdominal fistula, GI perforation, or intraabdominal abscess within 28 days prior to enrollment
* Previous major surgery within 28 days prior to enrollment
* Poorly controlled hypertension (defined as systolic blood pressure of ≥150 mmHg or diastolic blood pressure of >100 mmHg based on a mean of three measurements at approximately 2-minute intervals) NOTE: Initiation or adjustment of antihypertensive medication(s) is permitted within 30 days prior to enrollment.
* Known active infection requiring IV or oral anti-infective treatment
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal or cardiac disease)
* Subjects with brain metastases of non-CNS primary tumor are excluded if brain metastases are symptomatic and treated (surgery, radiation therapy) but not clinically and radiographically stable one month after local therapy (as assessed by contrast enhanced MRI or CT), OR asymptomatic and untreated but >1 cm in the longest dimension NOTE: Subjects with small (less than or equal to 1 cm in the longest dimension), asymptomatic brain metastases who do not need immediate local therapy may be enrolled.

NOTE: Subjects receiving a stable (i.e., unchanged) dose of corticosteroids for >30 days or subjects who have not received corticosteroids within 14 days prior to the first dose of study treatment may be enrolled. Subjects must not have received enzyme-inducing anticonvulsants within 28 days prior to enrollment.

* History or evidence of cardiovascular risk including any of the following: QTcF greater than or equal to 470 msec NOTE: If first screening QTcF is greater than or equal to 470 msec, ECG should be repeated two additional times at least five minutes apart and the average of the three readings should be used to determine eligibility. Clinically significant ECG abnormalities including second degree (Type II) or third degree AV block, history of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, stenting, or bypass grafting within the past six months prior to enrollment, Class III or IV heart failure as defined by the NYHA functional classification system, Left ventricular ejection fraction (LVEF) below the institutional LLN, NOTE: If a LLN does not exist at an institution, then use LVEF <50%, Baseline cTnI >10% CV, NTproBNP greater than or equal to 300 pg/mL, Known cardiac metastases
* Known hypersensitivity to any of the components of GSK2636771.
* For Tumor-Specific Expansion Cohort: CRC and Signal-finding Expansion Cohorts only: Female subjects who are pregnant, lactating or actively breastfeeding
* Known or active: Hepatitis B surface antigen or Hepatitis C antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-11-10 (Actual); Primary Completion 2015-11-12 (Actual); Study Completion 2016-02-25 (Actual)

PRIMARY OUTCOMES:
Part 1 (Initial Dose Selection): characterize safety, tolerability, and pharmacokinetics following single dose oral administration of GSK2636771 and to determine the starting dose for Part 2. | Single Dose Day 1 though 4
  Pharmacokinetic parameters including AUC, Cmax, tmax, and t1/2; adverse events, serious adverse events, changes in laboratory values, ECG parameters, and vital signs; median and maximum AUC(0-24)
Part 2 (Dose Escalation): characterize safety, tolerability, and pharmacokinetics following single- and repeat-dose oral administration of GSK2636771 and to determine the recommended dose and schedule for Part 3. | 4 weeks
  Pharmacokinetic parameters including AUC, Cmax, tmax, and t1/2; adverse events, serious adverse events, changes in laboratory values, ECG parameters, and vital signs; dose-limiting toxicities and/or biological activity in tumor or anti-tumor efficacy
Part 3 (Expansion cohorts):To further evaluate the clinical activity of oral GSK2636771 in PTEN deficient CRPC, CRC and multiple PTEN deficient tumor types. | Every 8 weeks
  Overall Response Rate (ORR): defined as the percentage of subjects with a confirmed complete response (CR) or partial response (PR) as per RECIST 1.1 criteria

SECONDARY OUTCOMES:
Part 1: characterize safety, tolerability, and pharmacokinetics following repeat-dose oral administration of GSK2636771. | Through 2 years
  adverse events, serious adverse events, changes in laboratory values, ECG parameters, and vital signs
Part 2: evaluate the pharmacodynamic (PD) response in PTEN deficient tumors after treatment with GSK2636771. | Through 2 years
  change from baseline in PD biomarkers which may include: platelet function, pathway proteins in tumor biopsy specimens and surrogate tissue, and/or soluble or cellular markers found in blood; ORR, defined as the percentage of subjects with a confirmed CR or PR as per RECIST 1.1 criteria; Duration of Response: defined, for the subset of subjects with a confirmed CR or PR, as the time from first documented evidence of CR or PR until first documented disease progression or death due to any cause
Part 3: further evaluate: the PD response in PTEN deficient tumors after treatment with GSK2636771; relationships between GSK2636771 PK, PD markers, and clinical endpoints; clinical tumor response after treatment with GSK2636771. | Through 2 years
  change from baseline in PD biomarkers which may include: platelet function, pathway proteins in tumor biopsy specimens/surrogate tissue, and/or soluble or cellular markers found in blood; change from baseline in circulating tumor cells (CTC) concentration in prostate cancer subjects; CTC Response Rate: defined as the number of subjects going from >5 CTCs to <5 CTCs per 7.5ml of blood (prostate cancer subjects only); Duration of Response; Progression Free Survival: defined as interval between date of first dose and earliest date of disease progression or death due to any cause
Part 3: further characterize the PK of GSK2636771, given orally, following single- and repeat-dose administration. | Through Day 23
  population pharmacokinetic parameters for GSK2636771 following single- and repeat-dose oral administration, including AUC and Vdss, and absorption rate constant (ka)
Part 3: further characterize the safety and tolerability of GSK2636771, given orally, following single- and repeat-dose administration. | Through 2 years
  adverse events and changes in laboratory values, ECG parameters, and vital signs following repeat-dose oral administration of GSK2636771
Part 3: confirm the Part 3 dose as the recommended Phase II dose (RP2D). | Through 2 years
  evaluation of all Part 3 measures

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (4):
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Salt Lake City, Utah
- GSK Investigational Site, Seoul, South Korea
- United Kingdom (2):
  - GSK Investigational Site, Sutton, Surrey
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: Results for study 115717 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115717?search=study&b'study_ids=115717'#rs